CLINICAL TRIAL: NCT05043740
Title: Effect of PCSK9 Inhibitor on Acute Coronary Syndrome Patients With Multivessel Disease and Relatively Low LDL-C Level in Chinese Population (CHOICE Study)
Brief Title: PCSK9 Inhibitor on ACS Patients With Multivessel Disease and Relatively Low LDL-C Level in Chinese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Shenghua Zhou, Director, Head of cardiovascular department, Principal Investigator, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHOICE202101
Record Dates: First submitted 2021-08-29; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — evolocumab; alirocumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care: management as recommended in ESC/EAS 2019 guidelines, within reimbursement criteria
- treatment (Experimental): On top of Standard of care, Evolocumab (Repatha®) 140 mg or Alirocumab(Praluent) 75mg every two weeks: first subcutaneous injection at the time of randomization, followings during 12 months.
  Interventions: Drug: Repatha or Praluent

INTERVENTIONS:
Drug: Repatha or Praluent — Evolocumab (Repatha®) 140 mg or Alirocumab (Praluent) 75mg every two weeks, first subcutaneous injection at the time of randomization, followings during 12 months
  Other Names: Evolocumab or Alirocumab
  Arms: treatment

SUMMARY:
The study is an open-label, multicenter, and randomized study. The objective of this study is to demonstrate the effect of PCSK9 inhibitor on ACS patients with multivessel disease and relatively low LDL-C levels or LDL-C levels lower than the recommended target.

The primary outcome was the rate of major adverse cardiac events (CV death, non-fatal myocardial infarction, documented unstable angina that requires admission into a hospital, all coronary revascularization with either PCI or CABG occurring at least 30 days after randomization, Non-fatal stroke) at 1 year. The secondary efficacy endpoints were individual components of the major adverse cardiac events, all cause death, and the percent change in LDL-C, Apo B, HDL-C, Lp(a) after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 40-85 years age;
* Recent hospitalization for acute coronary syndrome
* LDL-C ≤70 mg/dL (≤1.8 mmol/L) in patients who have been receiving stable treatment with moderate- or high-intensity statin within ≥ 4 weeks prior to enrollment (i.e. continuous treatment that has not changed with regard to statin intensity over the past 4 weeks) or, LDL-C ≤90 mg/dL (≤2.3 mmol/L) in patients who have been receiving stable treatment with low-intensity statin within ≥ 4 weeks prior to enrollment (i.e. continuous treatment that has not changed with regard to statin intensity over the past 4 weeks), or LDL-C≤125 mg/dL (≤3.2 mmol/L) in patients who are statin-naïve or have not been on a stable (unchanged) statin regimen for at least 4 weeks prior to enrollment;
* Multivessel disease, defined as ≥50% reduction in lumen diameter of at least three major epicardial coronary arteries by angiographic visual estimation or in major branches of one or more of these arteries, irrespective of the localization (proximal 50mm or more distal localization) of the obstructive lesions
* Patients with written informed consent.

Exclusion Criteria:

* Unstable clinical status (hemodynamic or electrical instability); Uncontrolled cardiac arrhythmia, defined as recurrent and symptomatic ventricular tachycardia or atrial fibrillation with rapid ventricular response not controlled by medications in the past 3 months prior to screening;
* Severe renal dysfunction, defined by estimated glomerular filtration rate <30 ml/min/1.73m2;
* Active liver disease or hepatic dysfunction, either reported in patient medical record or defined by asparate aminotransferase (AST) or alanine aminotransferase (ALT) levels > 3x the upper limit of normal;
* Patients who previously received evolocumab or other PCSK9 inhibitor;
* Treatment with systemic steroids or systemic cyclosporine in the past 3 months systemic cyclosporine, systemic steroids (eg. intravenous, intramuscular or per os);
* Known active infection or major hematologic, metabolic, or endocrine dysfunction in the judgment of the Investigator;
* Patients who will not be available for study-required procedures in the judgment of the Investigator;
* Current enrollment in another investigational device or drug study;
* Active malignancy requiring treatment;
* Intolerance of or allergy to statin or PCSK9 inhibitor;
* pregnancy, giving birth within the last 90 days, or lactation.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1360 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 12 months
  The primary endpoint in the CHOICE study was the rate of major adverse cardiac events at 1 year. The definition of major adverse cardiac events was a composite of:
  * CV death
  * Major coronary events 1) non-fatal myocardial infarction [MI]; 2)documented unstable angina that requires admission into a hospital; 3)all coronary revascularization with either PCI or CABG occurring at least 30 days after randomization)
  * Non-fatal stroke

SECONDARY OUTCOMES:
Secondary Endpoint | 12 months
  The secondary efficacy endpoints were individual components of the major adverse cardiac events, all cause death, and the percent change in LDL-C, Apo B, HDL-C, Lp(a) at 1 year.
Secondary Endpoint | 12 months
  the percent change in LDL-C, Apo B, HDL-C, Lp(a) at 1 year.